CLINICAL TRIAL: NCT00401518
Title: The Investigational Plan for the Evaluation of the ACADIA® Facet Replacement System
Brief Title: A Pivotal Study of a Facet Replacement System to Treat Spinal Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1020-9052
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Spinal Stenosis; Lumbar Spinal Stenosis; Facet Arthroplasty; Posterior Fusion; Facet Arthritis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACADIA® (Experimental): Investigational surgical treatment using the ACADIA Facet Replacement system
  Interventions: Device: Non-randomized ACADIA® Facet Replacement System; Device: Randomized ACADIA® Facet Replacement System
- Control Instrumented PLF (Active Comparator): Control surgical treatment using an instrumented posterolateral fusion
  Interventions: Device: Randomized Instrumented posterolateral fusion (PLF)

INTERVENTIONS:
Device: Non-randomized ACADIA® Facet Replacement System — Non-randomized investigational ACADIA Facet Replacement System used for the treatment of lumbar spinal stenosis
  Arms: ACADIA®
Device: Randomized ACADIA® Facet Replacement System — Randomized investigational ACADIA Facet Replacement System used for the treatment of lumbar spinal stenosis
  Arms: ACADIA®
Device: Randomized Instrumented posterolateral fusion (PLF) — Randomized control treatment using an instrumented posterolateral fusion for the treatment of lumbar spinal stenosis
  Arms: Control Instrumented PLF

SUMMARY:
The purpose of this study is to determine if the ACADIA® Facet Replacement System is effective in the treatment of spinal stenosis. The primary objective of the study is to evaluate the overall success rate of the Anatomic Facet Replacement System in patients with spinal stenosis when compared to a posterior spinal fusion control.

DETAILED DESCRIPTION:
Spinal Stenosis continues to be a major cause of back and leg pain. The condition is attributed to narrowing of the space around the nerves in the lumbar spine. This is often caused by the degenerative process in the spine and the facet joints. The current treatment calls for removal of bone around the affected nerve including the facet joints and fusing the posterior of the spine to ensure the segments remain stable.

The ACADIA® Facet Replacement System (AFRS) allows for an anatomic reconstruction of the facet joint after decompression and removal of the degenerated facet. Like the original facet joint, the replacement implant is designed to reproduce facet motion while restoring normal stability and motion.

The ACADIA® Facet Replacement System (AFRS) has been designed on the principals that have allowed other total joint replacement procedures to provide significant patient benefits. These guiding principals include:

* Anatomically based implant design
* Reproducible surgical technique
* Elimination of pain

The ACADIA® Facet Replacement System allows the surgeon to remove the offending bone while preserving the motion of the facet joint.

This study will evaluate the outcomes of patients using the AFRS™ investigation compared to those receiving instrumented posterior fusion procedure. Patients will be required to complete study visits before the procedure and at 6 weeks, 3, 6, 12, 24 months post procedure and annually thereafter as required by FDA. Follow up visits consist of administration of questionnaires, radiographs and neurological assessment.

ELIGIBILITY:
Inclusion Criteria:

* 21-85 years of age and skeletally mature;
* Have undergone 6 months of non-operative treatment prior to surgery;
* Lateral, lateral recess and/or central canal stenosis;
* Disc height measuring ≥ 4 mm at the operative level;
* Persistent leg, thigh and/or buttock symptoms,including pain,numbness, burning or tingling with a minimum leg pain score of 40mm as measured with the Visual Analogue Scale (VAS) Index;
* A score greater than 2 on a scale of 1-5 on the Zurich Claudication Questionnaire (ZCQ) Symptom Severity (SS) Score-Candidate;
* A score greater than or equal to 2 on a scale of 1-4 on the ZCQ Physical Function (PF) Score;
* A candidate for a decompression with full facetectomy at the operative level
* Candidate for a posterior lumbar fusion;
* Physically and mentally willing and able to comply evaluations;
* Lives in the immediate area and has no plans to relocate;

Exclusion Criteria:

* Previous surgical procedure at the operative or adjacent level except for one of the following: Micro-discectomy, laminectomy, lamino/foraminotomy, rhizotomy, IDET, and/or interspinous spacer;
* Previous lumbar fusion or disc replacement procedure;
* Osteoporosis;
* greater than Grade I spondylolisthesis or retrolisthesis;
* Spondylolisthesis at levels other than at the operative level;
* Scoliosis of the lumbar spine (defined as more than 11 deg Cobb angle) as indicated by plain X-ray films;
* Primary diagnosis of discogenic back pain due to torn, herniated, inflamed or irritated disc or other pathology where the patient exhibits axial back pain from degenerative disc disease;
* Acute traumatic pars fracture at the operative/adjacent level vertebral body;
* Spinal stenosis at more than three lumbar segments;
* Acute trauma to the lumbar spine within the last 24 months;
* Active infection at the operative level, or a systemic infection;
* Physically / mentally compromised;
* Systemic disease that would affect the patient's welfare or the research study.
* Immunologically suppressed or immunocompromised;
* Insulin-Dependent Diabetes Mellitus (Type I Diabetes);
* Currently undergoing long-term steroid therapy;
* Metabolic bone disease;
* Active malignancy: (except non-melanoma skin cancer), unless treated with no clinical signs or symptoms of the malignancy for at least 5 years;
* Known allergy to cobalt chromium or titanium;
* Used any investigational drug or device within the past 30 days;
* Pending litigation related to back pain or injury;
* Is a prisoner.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-10; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (28):
  - Spine Group Beverly Hills, Beverly Hills, California
  - Cedars-Sinai Spine Center, Los Angeles, California
  - Desert Orthopaedic Center, Rancho Mirage, California
  - Boulder Neurosurgical & Spine Associates, Boulder, Colorado
  - Spine Colorado, Durango, Colorado
  - Rocky Mountain Associates (RMA) in Orthopedic Medicine, Loveland, Colorado
  - Florida Spine Institute, Clearwater, Florida
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Neurological Institute of Savannah and Center for Spine, Savannah, Georgia
  - Indiana Spine Group, Carmel, Indiana
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Rubin Institute for Advanced Orthopaedics, Owings Mills, Maryland
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Spine Midwest, Inc., Jefferson City, Missouri
  - Springfield Neurological & Spine Institute, Springfield, Missouri
  - Albany Medical Center, Albany, New York
  - Carolina Neurosurgery and Spine Associates, P.C., Charlotte, North Carolina
  - OrthoCarolina Spine Center, Charlotte, North Carolina
  - Riverhills Healthcare, Cincinnati, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Charleston Brain & Spine, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Neuro-Spine Solutions, Bristol, Tennessee
  - The Center for Sports Medicine & Orthopedics, Chattanooga, Tennessee
  - Central Texas Spine Institute, Austin, Texas
  - University of Utah, Salt Lake City, Utah
- University of Puerto Rico, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-randomized ACADIA®: Non-randomized investigational surgical treatment using the ACADIA Facet Replacement system for the treatment of lumbar spinal stenosis
- Randomized ACADIA®: Randomized investigational surgical treatment using the ACADIA Facet Replacement system for the treatment of lumbar spinal stenosis
- Randomized Instrumented PLF: Randomized control surgical treatment using an instrumented posterolateral fusion for the treatment of lumbar spinal stenosis
Period: Overall Study
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Started | 46 | 227 | 117
Completed | 40 | 190 | 94
Not Completed | 6 | 37 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF | Total
Number analyzed (Participants) | 46 | 227 | 117 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (11.46) | 61.7 (9.82) | 61.4 (10.55) | 61.2 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 119 | 55 | 196
  Male | 24 | 108 | 62 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 0 | 5 | 0 | 5
  Black or African American | 1 | 2 | 7 | 10
  Caucasian | 41 | 206 | 103 | 350
  Hispanic | 3 | 12 | 7 | 22
  Other | 1 | 2 | 0 | 3
Height [Mean (Standard Deviation); unit: inches] | 67.3 (3.91) | 66.9 (4.41) | 67.4 (3.86) | 67.1 (4.19)
Weight [Mean (Standard Deviation); unit: pounds] | 190.8 (41.34) | 191.3 (39.62) | 191.2 (37.38) | 191.2 (39.07)

OUTCOME MEASURES:

1. Primary Outcome: Measure of Pain/Disability Using the Zurich Claudication Questionnaire (ZCQ) Physical Function Score
Description: Physical Function is measured on a scale of 1-4 points (lower values are considered a better outcome)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 40 | 190 | 94
score on a scale | 1.7 (0.71) | 1.6 (0.62) | 1.7 (0.73)

2. Primary Outcome: Measure of Pain/Disability Using the Zurich Claudication Questionnaire (ZCQ) Symptom Severity Score
Description: Symptom Severity is measured on a scale of 1-5 points (lower values are considered a better outcome)
Time Frame: 24 months
Population: One patient from the Randomized ACADIA group did not have ZCQ Symptom Severity data at 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 40 | 189 | 94
score on a scale | 2.1 (0.90) | 2.0 (0.80) | 2.2 (0.98)

3. Primary Outcome: Number of Participants Who Maintained or Improved in Neurological Status.
Description: Neurological status is based on four types of measurement parameters: muscle strength, straight leg raise, sensory function, and reflexes. Each of the four parameters will be coded as Stable or Improved OR Deteriorated. Neurological assessment scores must be stable or improved compared with the preoperative baseline to be considered "Stable or Improved" neurological status. If these scores have deteriorated as compared to the preoperative baseline, then the neurological status is considered "Deteriorated".
Time Frame: 24 months
Population: Only patients with Neurological data at 24 months and treated with ACADIA or the control treatment were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 43 | 204 | 99
Participants | 30 | 155 | 75

4. Secondary Outcome: Mean Visual Analog Scale (VAS) Right Leg Pain
Description: The visual analog scale (VAS) is a questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "as severe as it could be" on the right border. The subject is instructed to make a mark along the line to represent the intensity of right leg pain currently being experienced; 0mm is equal to no pain and 100mm is pain as severe as it could be. The clinician records the distance of the mark in millimeters from the left end of the scale.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 40 | 190 | 94
score on a scale | 19.4 (28.11) | 13.2 (24.97) | 22.5 (30.80)

5. Secondary Outcome: Mean Visual Analog Scale (VAS) Left Leg Pain
Description: The visual analog scale (VAS) is a questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "as severe as it could be" on the right border. The subject is instructed to make a mark along the line to represent the intensity of left leg pain currently being experienced; 0mm is equal to no pain and 100mm is pain as severe as it could be. The clinician records the distance of the mark in millimeters from the left end of the scale.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 40 | 190 | 94
score on a scale | 17.5 (29.72) | 12.2 (24.25) | 16.9 (26.68)

6. Secondary Outcome: Mean Visual Analog Scale (VAS) Back Pain
Description: The visual analog scale (VAS) is a questionnaire used to quantify a subjective experience, such as the intensity of pain. The scale is a 100mm line labeled with "no pain" on the left border and "as severe as it could be" on the right border. The subject is instructed to make a mark along the line to represent the intensity of back pain currently being experienced; 0mm is equal to no pain and 100mm is pain as severe as it could be. The clinician records the distance of the mark in millimeters from the left end of the scale.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 40 | 190 | 94
score on a scale | 24.7 (30.23) | 18.8 (25.24) | 23.9 (26.86)

7. Secondary Outcome: Number of Participants With a Change of at Least 15 Points in Pain/Disability Using the Oswestry Disability Index (ODI) Score at 24 Months Compared With the Score at Baseline
Description: The Oswestry Disability Index (ODI) is a commonly used outcome-measure questionnaire for low back pain in a hospital setting. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Time Frame: 24 months
Population: Six Non-randomized ACADIA®, 37 Randomized ACADIA® and 23 Randomized instrumented PLF did not complete the 24 month visit and thus were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
Number analyzed (Participants) | 40 | 190 | 94
Participants | 33 | 151 | 62

ADVERSE EVENTS:
Time Frame: 24 months
Description: The Total Number of Participants at Risk for the "Randomized ACADIA" Arm/Group is not consistent with numbers provided in the Participant Flow module. The discrepancy is due to one patient being randomized to ACADIA but not receiving the ACADIA treatment. This patient is included in the intent-to-treat population for efficacy analyses. It is not possible to make any changes to data including Adverse Event Terms as the study is closed and all analysis is complete.
Arm/Group | Non-randomized ACADIA® | Randomized ACADIA® | Randomized Instrumented PLF
All-Cause Mortality (participants affected / at risk) | 2/46 | 4/226 | 3/117
Serious Adverse Events (participants affected / at risk) | 20/46 | 111/226 | 40/117
Other Adverse Events (participants affected / at risk) | 46/46 | 213/226 | 108/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized ACADIA® (N=46) | Randomized ACADIA® (N=226) | Randomized Instrumented PLF (N=117)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5 | 0
Cardiovascular (Cardiac disorders) | 3 | 15 | 7
Death (General disorders) | 0 | 4 | 0
Gastrointestinal (Gastrointestinal disorders) | 3 | 12 | 6
Infection - Deep Wound (Infections and infestations) | 0 | 3 | 0
Other (General disorders) | 0 | 5 | 2
Psychological (Psychiatric disorders) | 0 | 1 | 0
Trauma (General disorders) | 2 | 1 | 3
Urogenital (Renal and urinary disorders) | 4 | 5 | 2
Infection - Other (Infections and infestations) | 2 | 8 | 5
Infection - Superficial Wound (Infections and infestations) | 0 | 1 | 0
Cerebrovascular (Vascular disorders) | 0 | 5 | 1
Surgery - Adjacent Level (Surgical and medical procedures) | 1 | 10 | 0
Wound Issue (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 5
Vertebral Fracture (General disorders) | 0 | 1 | 0
Pain-Neck and/or Upper Extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Pain-Back and Lower Extremities (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain Lower Extremities (Musculoskeletal and connective tissue disorders) | 2 | 13 | 8
Pain - Hip (Musculoskeletal and connective tissue disorders) | 1 | 11 | 2
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Surgery - Index Level (Surgical and medical procedures) | 7 | 35 | 13
Surgery - Other (Non-Lumbar) (Surgical and medical procedures) | 1 | 1 | 0
Surgery - Other Lumbar (Surgical and medical procedures) | 1 | 0 | 1
Dural Tear (Nervous system disorders) | 0 | 2 | 1
Neurological Focal Lumbar (Nervous system disorders) | 0 | 1 | 0
Radiographic (General disorders) | 0 | 1 | 0
Metal Allergy (Immune system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized ACADIA® (N=46) | Randomized ACADIA® (N=226) | Randomized Instrumented PLF (N=117)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 4
Cardiovascular (Cardiac disorders) | 10 | 21 | 13
Dysesthesia - Upper Extremities (Nervous system disorders) | 1 | 0 | 1
Gastrointestinal (Gastrointestinal disorders) | 9 | 32 | 9
Headache (General disorders) | 1 | 3 | 0
Other (General disorders) | 20 | 42 | 24
Pain - Other (General disorders) | 0 | 5 | 2
Psychological (Psychiatric disorders) | 0 | 8 | 1
Trauma (General disorders) | 11 | 42 | 26
Urogenital (Renal and urinary disorders) | 2 | 21 | 5
Dysesthesia - Lower Extremities (Nervous system disorders) | 2 | 2 | 2
Infection - Superficial Wound (Infections and infestations) | 1 | 4 | 2
Infection - Other (Infections and infestations) | 9 | 23 | 17
Cerebrovascular (Vascular disorders) | 1 | 3 | 0
Surgery - Adjacent Level (Surgical and medical procedures) | 0 | 3 | 2
Wound Issue (Skin and subcutaneous tissue disorders) | 1 | 5 | 4
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 | 16 | 7
Spinous Process Fracture (General disorders) | 0 | 1 | 0
Vertebral Fracture (General disorders) | 0 | 2 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Pain-Neck and/or Upper Extremity (Musculoskeletal and connective tissue disorders) | 9 | 30 | 22
Pain - Back (Musculoskeletal and connective tissue disorders) | 19 | 72 | 27
Pain-Back and Lower Extremities (Musculoskeletal and connective tissue disorders) | 6 | 34 | 17
Pain - Back and Hip (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Pain Lower Extremities (Musculoskeletal and connective tissue disorders) | 18 | 68 | 38
Pain - Hip (Musculoskeletal and connective tissue disorders) | 12 | 28 | 14
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 | 18 | 13
Neurological Systemic (Nervous system disorders) | 1 | 4 | 1
Dysesthesia - Other (Nervous system disorders) | 0 | 3 | 1
Pain-Back and Lower Extremities with Dysesthesia (Musculoskeletal and connective tissue disorders) | 2 | 10 | 2
Pain-Back with Dysesthesia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Pain Lower Extremities with Dysesthesia (Musculoskeletal and connective tissue disorders) | 3 | 8 | 5
Surgery-Index Level (Surgical and medical procedures) | 2 | 6 | 1
Surgery - Other (Non-Lumbar) (Surgical and medical procedures) | 1 | 2 | 0
Weakness (General disorders) | 0 | 2 | 4
Paresthesia - Upper Extremities (Nervous system disorders) | 4 | 7 | 4
Paresthesia - Lower Extremities (Nervous system disorders) | 4 | 22 | 10
Paresthesia - Other (Nervous system disorders) | 1 | 0 | 0
Pseudoarthrosis (Hepatobiliary disorders) | 0 | 0 | 2
Surgery - Other Lumbar (Surgical and medical procedures) | 0 | 1 | 0
Dural Tear (General disorders) | 2 | 22 | 12
Neurological Focal Lumbar (Nervous system disorders) | 21 | 104 | 50
Neurolgical Focal Other (Nervous system disorders) | 3 | 10 | 3
Peripheral Neuropathy (Nervous system disorders) | 1 | 5 | 1
Radiographic (General disorders) | 1 | 5 | 0
Metal Allergy (Immune system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To prevent premature disclosure of trade secrets or other confidential information, Investigator agrees not to present, publish, or disclose study results or information about the investigational device without the express written consent of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT00401518/Prot_SAP_000.pdf